CLINICAL TRIAL: NCT02987972
Title: A Phase II, Double-Blind, Randomized, Multicenter Trial to Evaluate the Safety, Tolerability, and Immunogenicity of V114 Compared to Prevnar 13™ in Healthy Infants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of Two Lots of V114 in Healthy Infants (V114-008)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: V114-008; 2016-001117-25 (EudraCT Number)
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-09

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- V114 Lot 1 (Experimental): Infants will receive a 0.5 mL intramuscular injection of V114 Lot 1 at 2, 4, 6, and 12-15 months of age (Study Day 1, Month 2, Month 4, and Month 10-13)
  Interventions: Biological: V114 Lot 1
- V114 Lot 2 (Experimental): Infants will receive a 0.5 mL intramuscular injection of V114 Lot 2 at 2, 4, 6, and 12-15 months of age (Study Day 1, Month 2, Month 4, and Month 10-13)
  Interventions: Biological: V114 Lot 2
- Prevnar 13™ (Active Comparator): Infants will receive a 0.5 mL intramuscular injection of Prevnar 13™ at 2, 4, 6, and 12-15 months of age (Study Day 1, Month 2, Month 4, and Month 10-13)
  Interventions: Biological: Prevnar 13™

INTERVENTIONS:
Biological: V114 Lot 1 — Lot 1: Pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, 33F (2 mcg each), and serotype 6B (4 mcg) in each 0.5 mL dose
  Other Names: V114-1
  Arms: V114 Lot 1
Biological: V114 Lot 2 — Lot 2: Pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19F, 19A, 22F, 23F, 33F (2 mcg each), and serotype 6B (4 mcg) in each 0.5 mL dose
  Other Names: V114-2
  Arms: V114 Lot 2
Biological: Prevnar 13™ — Pneumococcal capsular polysaccharide serotypes 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 23F (2.2 mcg) and 6B (4.4 mcg) in each 0.5 ml dose
  Arms: Prevnar 13™

SUMMARY:
This study is designed to evaluate the safety, tolerability, and immunogenicity of two different lots of V114 in healthy infants 6 to 12 weeks (>=42 days to <=90 days) of age. The primary hypothesis of the study is that the proportion of participants receiving V114 who have serotype specific IgG >=0.35 mcg/mL for each of pneumococcal serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F at 1 month after Dose 3 is non-inferior to that for recipients of Prevnar 13™.

ELIGIBILITY:
Inclusion Criteria:

* Infant approximately 2 months of age (42 days to 90 days), inclusive
* In good health

Exclusion Criteria:

* Prior administration of any pneumococcal vaccine
* Known hypersensitivity to any component of the pneumococcal conjugate vaccine or any diphtheria toxoid-containing vaccine
* Known or suspected impairment of immunological function
* History of congenital or acquired immunodeficiency (eg, splenomegaly)
* Mother has documented human immunodeficiency virus (HIV) infection
* Mother has documented hepatitis B surface antigen-positive test result
* Known or history of functional or anatomic asplenia
* History of failure to thrive
* History of a coagulation disorder
* History of autoimmune disease
* Known neurologic or cognitive behavioral disorder
* Expects to require systemic corticosteroids within 30 days after each vaccination during the trial
* Prior administration of a blood transfusion or blood products, including immunoglobulin
* Participated in another clinical trial of an investigational product
* History of invasive pneumococcal disease or known history of other culture-positive pneumococcal disease

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1051 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (49):
- United States (30):
  - Birmingham Pediatric Research ( Site 0043), Birmingham, Alabama
  - Southeastern Pediatric Associates, P.A. ( Site 0079), Dothan, Alabama
  - Children's Clinic of Jonesboro, PA ( Site 0054), Jonesboro, Arkansas
  - Premier Health Research Center, LLC ( Site 0035), Downey, California
  - Sherif Khamis MD, Inc. ( Site 0044), Palmdale, California
  - Kaiser Permanente - Roseville ( Site 0045), Roseville, California
  - Kaiser Permanente Clinical Trial - Sacramento ( Site 0076), Sacramento, California
  - Kentucky Pediatric/Adult Research Inc ( Site 0037), Bardstown, Kentucky
  - University of Louisville: Pediatric Clinical Trials Unit ( Site 0049), Louisville, Kentucky
  - ACC Pediatric Research ( Site 0039), Haughton, Louisiana
  - Woburn Pediatric Associates ( Site 0046), Woburn, Massachusetts
  - Dundee Clinic ( Site 0063), Omaha, Nebraska
  - Child Health Care Associates ( Site 0064), East Syracuse, New York
  - State University of New York Upstate Medical University ( Site 0065), Syracuse, New York
  - Pediatric Associates of Mt. Carmel, Inc. ( Site 0052), Cincinnati, Ohio
  - Senders Pediatrics ( Site 0058), Cleveland, Ohio
  - Ohio Pediatric Research Association ( Site 0060), Dayton, Ohio
  - Pediatric Medical Associates ( Site 0059), East Norriton, Pennsylvania
  - Kid's Way Pediatrics ( Site 0036), Hermitage, Pennsylvania
  - Thomas Jefferson University ( Site 0067), Philadelphia, Pennsylvania
  - Coastal Pediatric Research ( Site 0070), Charleston, South Carolina
  - Holston Medical Group [Kingsport, TN] ( Site 0048), Kingsport, Tennessee
  - University of Texas Medical Branch at Galveston ( Site 0056), Galveston, Texas
  - University of Texas Medical Branch at Galveston ( Site 0068), League City, Texas
  - Wee Care Pediatrics ( Site 0042), Layton, Utah
  - Cottonwood Pediatrics ( Site 0041), Murray, Utah
  - Copperview Medical Center ( Site 0062), South Jordan, Utah
  - Pediatric Research of Charlottesville, LLC ( Site 0066), Charlottesville, Virginia
  - Huguenot Pediatrics ( Site 0057), Midlothian, Virginia
  - Family Health Care of Ellensburg ( Site 0077), Ellensburg, Washington
- Canada (3):
  - CHU Ste-Justine ( Site 0084), Montreal, Quebec
  - McGill University Health Centre - Vaccine Study Centre ( Site 0030), Pierrefonds, Quebec
  - CHU de Quebec Universite de Laval ( Site 0031), Québec, Quebec
- Denmark (2):
  - Aarhus Universitetshospital-Skejby-Forskningsklinikken for Kvindesygdomme ( Site 0025), Aarhus N
  - OUH Klinisk Forsk center Gyn Obs D. ( Site 0024), Odense
- Finland (8):
  - Tampereen yliopisto Espoon rokotetutkimusklinikka ( Site 0007), Espoo
  - Tampereen yliopisto Etela-Helsingin rokotetutkimusklinikka ( Site 0005), Helsinki
  - Tampereen yliopisto Ita-Helsingin rokotetutkimusklinikka ( Site 0006), Helsinki
  - Tampereen yliopisto Järvenpään rokotetutkimusklinikka ( Site 0003), Jarvenpaa
  - Tampereen yliopisto Oulun rokotetutkimusklinikka ( Site 0004), Oulu
  - Tampereen yliopisto Porin rokotetutkimusklinikka ( Site 0008), Pori
  - Tampereen yliopisto - Tampereen rokotetutkimusklinikka ( Site 0001), Tampere
  - Tampereen yliopisto Turun rokotetutkimusklinikka ( Site 0002), Turku
- Israel (4):
  - Soroka University Medical Center ( Site 0019), Beersheba
  - Soroka University Medical Center - Rahat Family health center ( Site 0020), Beersheba
  - Soroka University Medical Center - Ramot Family health center ( Site 0021), Beersheba
  - Soroka University Medical Center - Vav Family health center ( Site 0022), Beersheba
- Spain (2):
  - Hospital Clinico Universitario de Santiago ( Site 0016), Santiago de Compostela
  - Unidad de Estudios e Investigacion IHP ( Site 0017), Seville

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Platt HL, Greenberg D, Tapiero B, Clifford RA, Klein NP, Hurley DC, Shekar T, Li J, Hurtado K, Su SC, Nolan KM, Acosta CJ, McFetridge RD, Bickham K, Musey LK; V114-008 Study Group. A Phase II Trial of Safety, Tolerability and Immunogenicity of V114, a 15-Valent Pneumococcal Conjugate Vaccine, Compared With 13-Valent Pneumococcal Conjugate Vaccine in Healthy Infants. Pediatr Infect Dis J. 2020 Aug;39(8):763-770. doi: 10.1097/INF.0000000000002765. PMID 32639460

RESULTS

PARTICIPANT FLOW:
Groups:
- V114 Lot 1: Infants received a 0.5 mL intramuscular injection of V114 Lot 1 at 2, 4, 6, and 12-15 months of age (Study Day 1, Month 2, Month 4, and Month 10-13)
- V114 Lot 2: Infants received a 0.5 mL intramuscular injection of V114 Lot 2 at 2, 4, 6, and 12-15 months of age (Study Day 1, Month 2, Month 4, and Month 10-13)
- Prevnar 13™: Infants received a 0.5 mL intramuscular injection of Prevnar 13™ at 2, 4, 6, and 12-15 months of age (Study Day 1, Month 2, Month 4, and Month 10-13)
Period: Overall Study
Arm/Group | V114 Lot 1 | V114 Lot 2 | Prevnar 13™
Started | 351 | 350 | 350
Vaccination 1 | 350 | 347 | 347
Vaccination 2 | 333 | 335 | 335
Vaccination 3 | 330 | 331 | 332
Vaccination 4 | 310 | 306 | 311
Completed | 308 | 305 | 308
Not Completed | 43 | 45 | 42
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lack of Efficacy | 9 | 12 | 12
Not completed — Lost to Follow-up | 7 | 8 | 4
Not completed — Physician Decision | 1 | 6 | 0
Not completed — Protocol Violation | 2 | 1 | 5
Not completed — Withdrawal by Subject | 22 | 17 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V114 Lot 1 | V114 Lot 2 | Prevnar 13™ | Total
Number analyzed (Participants) | 351 | 350 | 350 | 1051
Age, Customized [Count of Participants; unit: Participants]
  Infants and toddlers (28 days-23 months) | 351 | 350 | 350 | 1051
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 164 | 186 | 173 | 523
  Male | 187 | 164 | 177 | 528
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 1 | 2 | 6
  Asian | 3 | 1 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 1 | 6
  Black or African American | 34 | 24 | 33 | 91
  White | 290 | 296 | 289 | 875
  More than one race | 18 | 25 | 22 | 65
  Unknown or Not Reported | 0 | 1 | 0 | 1
Ethnicity [Count of Participants; unit: Participants]
  Hispanic Or Latino | 49 | 36 | 53 | 138
  Not Hispanic Or Latino | 300 | 313 | 294 | 907
  Not Reported | 0 | 0 | 2 | 2
  Unknown | 2 | 1 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving the Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody Threshold Value of ≥0.35 µg/mL for the 13 Common Serotypes in V114 and Prevnar 13™: 1 Month Post Vaccination 3
Description: Serotype-specific pneumococcal IgG antibody was measured using the Meso-Scale Discovery (MSD) Pneumococcal electrochemiluminescence assay (Pn ECL). The percentage of participants with serotype-specific IgG ≥0.35 µg/mL was summarized for each serotype.
Time Frame: 1 month post vaccination 3 (Month 5)
Population: Participants not considered as protocol violators and had data available for endpoint. Violations could include but were not limited to: failure to receive the scheduled correct doses within scheduled timeframe and lack of valid serology results available from 28 to 42 days following the dose being analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V114 Lot 1 | V114 Lot 2 | Prevnar 13™
Number analyzed (Participants) | 329 | 330 | 332
Percentage of Participants
  Type 1: number analyzed (Participants) | 278 | 273 | 291
  Type 1 | 96.8 [93.94 to 98.51] | 97.8 [95.28 to 99.19] | 96.9 [94.21 to 98.58]
  Type 3: number analyzed (Participants) | 277 | 273 | 291
  Type 3 | 96.0 [93.01 to 98.00] | 94.1 [90.66 to 96.61] | 71.8 [66.28 to 76.92]
  Type 4: number analyzed (Participants) | 273 | 272 | 288
  Type 4 | 98.2 [95.78 to 99.40] | 97.1 [94.29 to 98.72] | 95.1 [91.98 to 97.32]
  Type 5: number analyzed (Participants) | 278 | 272 | 290
  Type 5 | 96.0 [93.03 to 98.01] | 96.0 [92.88 to 97.96] | 96.6 [93.75 to 98.33]
  Type 6A: number analyzed (Participants) | 278 | 273 | 290
  Type 6A | 90.6 [86.60 to 93.80] | 95.6 [92.45 to 97.71] | 96.2 [93.31 to 98.09]
  Type 6B: number analyzed (Participants) | 276 | 273 | 290
  Type 6B | 90.6 [86.50 to 93.75] | 92.3 [88.48 to 95.18] | 91.4 [87.54 to 94.34]
  Type 7F: number analyzed (Participants) | 278 | 273 | 290
  Type 7F | 99.6 [98.01 to 99.99] | 99.3 [97.38 to 99.91] | 99.0 [97.01 to 99.79]
  Type 9V: number analyzed (Participants) | 278 | 273 | 289
  Type 9V | 97.1 [94.41 to 98.75] | 97.8 [95.28 to 99.19] | 95.8 [92.86 to 97.84]
  Type 14: number analyzed (Participants) | 277 | 273 | 289
  Type 14 | 99.3 [97.42 to 99.91] | 97.4 [94.79 to 98.96] | 97.2 [94.62 to 98.80]
  Type 18C: number analyzed (Participants) | 278 | 273 | 291
  Type 18C | 96.8 [93.94 to 98.51] | 98.2 [95.78 to 99.40] | 95.5 [92.48 to 97.60]
  Type 19A: number analyzed (Participants) | 278 | 273 | 290
  Type 19A | 98.9 [96.88 to 99.78] | 98.5 [96.29 to 99.60] | 98.6 [96.51 to 99.62]
  Type 19F: number analyzed (Participants) | 278 | 273 | 290
  Type 19F | 100.0 [98.68 to 100.00] | 98.9 [96.82 to 99.77] | 99.7 [98.09 to 99.99]
  Type 23F: number analyzed (Participants) | 278 | 273 | 290
  Type 23F | 92.4 [88.68 to 95.26] | 94.9 [91.55 to 97.17] | 90.7 [86.74 to 93.77]
Statistical Analysis 1: Comparison: V114 Lot 1 vs Prevnar 13™; Type 1; Test type: Non-Inferiority — Statistical criterion for non-inferiority corresponds to the lower bound of the adjusted 95% CI of the proportion difference (V114 minus Prevnar 13™) being greater than -0.15 for each of the 13 shared serotypes; p < 0.001, Miettinen and Nurminen; Difference in Percentages = -0.1, 95% CI 2-sided [-3.3 to 3.0] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 2: Comparison: V114 Lot 1 vs Prevnar 13™; Type 3; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 24.2, 95% CI 2-sided [18.7 to 30.0] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar
Statistical Analysis 3: Comparison: V114 Lot 1 vs Prevnar 13™; Type 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 3.0, 95% CI 2-sided [0.0 to 6.4] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 4: Comparison: V114 Lot 1 vs Prevnar 13™; Type 5; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = -0.5, 95% CI 2-sided [-3.9 to 2.8] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 5: Comparison: V114 Lot 1 vs Prevnar 13™; Type 6A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = -5.6, 95% CI 2-sided [-10.0 to -1.6] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 6: Comparison: V114 Lot 1 vs Prevnar 13™; Type 6B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = -0.8, 95% CI 2-sided [-5.7 to 4.0] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 7: Comparison: V114 Lot 1 vs Prevnar 13™; Type 7F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 0.7, 95% CI 2-sided [-1.1 to 2.7] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 8: Comparison: V114 Lot 1 vs Prevnar 13™; Type 9V; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 1.3, 95% CI 2-sided [-1.9 to 4.6] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 9: Comparison: V114 Lot 1 vs Prevnar 13™; Type 14; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 2.0, 95% CI 2-sided [-0.2 to 4.7] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 10: Comparison: V114 Lot 1 vs Prevnar 13™; Type 18C; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 1.2, 95% CI 2-sided [-2.1 to 4.7] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 11: Comparison: V114 Lot 1 vs Prevnar 13™; Type 19A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 0.3, 95% CI 2-sided [-1.9 to 2.6] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 12: Comparison: V114 Lot 1 vs Prevnar 13™; Type 19F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 0.3, 95% CI 2-sided [-1.0 to 1.9] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 13: Comparison: V114 Lot 1 vs Prevnar 13™; Type 23F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 1.8, 95% CI 2-sided [-2.9 to 6.5] — Difference in Response Rate calculated as Percentage V114 Lot 1 minus Percentage Prevnar 13™
Statistical Analysis 14: Comparison: V114 Lot 2 vs Prevnar 13™; Type 1; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 0.9, 95% CI 2-sided [-2.0 to 3.9] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 15: Comparison: V114 Lot 2 vs Prevnar 13™; Type 3; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 22.3, 95% CI 2-sided [16.5 to 28.3] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 16: Comparison: V114 Lot 2 vs Prevnar 13™; Type 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 1.9, 95% CI 2-sided [-1.4 to 5.4] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 17: Comparison: V114 Lot 2 vs Prevnar 13™; Type 5; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = -0.6, 95% CI 2-sided [-4.1 to 2.7] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 18: Comparison: V114 Lot 2 vs Prevnar 13™; Type 6A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = -0.6, 95% CI 2-sided [-4.2 to 2.8] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 19: Comparison: V114 Lot 2 vs Prevnar 13™; Type 6B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 0.9, 95% CI 2-sided [-3.7 to 5.6] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 20: Comparison: V114 Lot 2 vs Prevnar 13™; Type 7F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 0.3, 95% CI 2-sided [-1.7 to 2.4] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 21: Comparison: V114 Lot 2 vs Prevnar 13™; Type 9V; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 2.0, 95% CI 2-sided [-1.1 to 5.2] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 22: Comparison: V114 Lot 2 vs Prevnar 13™; Type 14; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 0.2, 95% CI 2-sided [-2.8 to 3.1] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 23: Comparison: V114 Lot 2 vs Prevnar 13™; Type 18C; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 2.6, 95% CI 2-sided [-0.3 to 5.9] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 24: Comparison: V114 Lot 2 vs Prevnar 13™; Type 19A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = -0.1, 95% CI 2-sided [-2.5 to 2.2] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 25: Comparison: V114 Lot 2 vs Prevnar 13™; Type 19F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = -0.8, 95% CI 2-sided [-2.9 to 0.9] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™
Statistical Analysis 26: Comparison: V114 Lot 2 vs Prevnar 13™; Type 23F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p < 0.001, Miettinen and Nurminen; Difference in Percentages = 4.2, 95% CI 2-sided [-0.1 to 8.7] — Difference in Response Rate calculated as Percentage V114 Lot 2 minus Percentage Prevnar 13™

2. Primary Outcome: Geometric Mean Concentration of Serotype-specific Pneumococcal IgG Antibody for the 13 Common Serotypes in V114 and Prevnar 13™ and the 2 Serotypes Unique to V114: 1 Month Post Vaccination 3
Description: Serotype-specific pneumococcal IgG antibody will be assayed using the Meso-Scale Discovery (MSD) Pn electrochemiluminescence assay. The geometric mean concentration (GMC) of serotype-specific IgG will be assessed.
Time Frame: 1 month post Vaccination 3 (Month 5)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 Lot 1 | V114 Lot 2 | Prevnar 13™
Number analyzed (Participants) | 329 | 330 | 332
µg/mL
  Type 1: number analyzed (Participants) | 278 | 273 | 291
  Type 1 | 1.19 [1.10 to 1.27] | 1.37 [1.26 to 1.49] | 1.65 [1.50 to 1.82]
  Type 3: number analyzed (Participants) | 277 | 273 | 291
  Type 3 | 1.04 [0.97 to 1.12] | 1.02 [0.93 to 1.11] | 0.53 [0.48 to 0.58]
  Type 4: number analyzed (Participants) | 273 | 272 | 288
  Type 4 | 1.30 [1.21 to 1.40] | 1.27 [1.17 to 1.37] | 1.26 [1.14 to 1.38]
  Type 5: number analyzed (Participants) | 278 | 272 | 290
  Type 5 | 1.37 [1.25 to 1.50] | 1.45 [1.32 to 1.59] | 1.75 [1.58 to 1.94]
  Type 6A: number analyzed (Participants) | 278 | 273 | 290
  Type 6A | 1.42 [1.27 to 1.59] | 1.48 [1.34 to 1.63] | 2.62 [2.35 to 2.92]
  Type 6B: number analyzed (Participants) | 276 | 273 | 290
  Type 6B | 1.95 [1.68 to 2.28] | 1.71 [1.49 to 1.96] | 1.89 [1.64 to 2.18]
  Type 7F: number analyzed (Participants) | 278 | 273 | 290
  Type 7F | 2.43 [2.26 to 2.62] | 2.42 [2.23 to 2.62] | 2.98 [2.72 to 3.26]
  Type 9V: number analyzed (Participants) | 278 | 273 | 289
  Type 9V | 1.40 [1.28 to 1.52] | 1.70 [1.56 to 1.86] | 1.59 [1.44 to 1.76]
  Type 14: number analyzed (Participants) | 277 | 273 | 289
  Type 14 | 5.08 [4.63 to 5.58] | 4.78 [4.27 to 5.34] | 5.79 [5.11 to 6.55]
  Type 18C: number analyzed (Participants) | 278 | 273 | 291
  Type 18C | 1.24 [1.15 to 1.35] | 1.65 [1.52 to 1.79] | 1.67 [1.52 to 1.82]
  Type 19A: number analyzed (Participants) | 278 | 273 | 290
  Type 19A | 1.63 [1.52 to 1.76] | 1.64 [1.51 to 1.78] | 1.99 [1.83 to 2.18]
  Type 19F: number analyzed (Participants) | 278 | 273 | 290
  Type 19F | 2.26 [2.10 to 2.43] | 2.33 [2.15 to 2.53] | 2.57 [2.38 to 2.78]
  Type 23F: number analyzed (Participants) | 278 | 273 | 290
  Type 23F | 1.22 [1.10 to 1.35] | 1.47 [1.32 to 1.63] | 1.25 [1.11 to 1.40]
  Type 22F: number analyzed (Participants) | 278 | 273 | 291
  Type 22F | 4.80 [4.40 to 5.24] | 4.18 [3.76 to 4.63] | 0.05 [0.05 to 0.06]
  Type 33F: number analyzed (Participants) | 278 | 273 | 289
  Type 33F | 1.58 [1.34 to 1.86] | 1.51 [1.30 to 1.75] | 0.05 [0.04 to 0.05]
Statistical Analysis 1: Comparison: V114 Lot 1 vs Prevnar 13™; Type 1; Test type: Other; GMC Ratio = 0.72, 95% CI 2-sided [0.64 to 0.81] — IgG GMC Ratio (V114 Lot 1/Prevnar 13™) based on analysis of variance (ANOVA) model with log-transformed IgG antibody responses as response variable and vaccination group as covariate
Statistical Analysis 2: Comparison: V114 Lot 1 vs Prevnar 13™; Type 3; Test type: Other; GMC Ratio = 1.98, 95% CI 2-sided [1.75 to 2.23] — IgG GMC Ratio (V114 Lot 1/Prevnar 13™) based on ANOVA model with log-transformed IgG antibody responses as response variable and vaccination group as covariate
Statistical Analysis 3: Comparison: V114 Lot 1 vs Prevnar 13™; Type 4; Test type: Other; GMC Ratio = 1.04, 95% CI 2-sided [0.92 to 1.16] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 4: Comparison: V114 Lot 1 vs Prevnar 13™; Type 5; Test type: Other; GMC Ratio = 0.78, 95% CI 2-sided [0.68 to 0.89] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 5: Comparison: V114 Lot 1 vs Prevnar 13™; Type 6A; Test type: Other; GMC Ratio = 0.54, 95% CI 2-sided [0.47 to 0.63] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 6: Comparison: V114 Lot 1 vs Prevnar 13™; Type 6B; Test type: Other; GMC Ratio = 1.03, 95% CI 2-sided [0.84 to 1.26] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 7: Comparison: V114 Lot 1 vs Prevnar 13™; Type 7F; Test type: Other; GMC Ratio = 0.82, 95% CI 2-sided [0.73 to 0.92] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 8: Comparison: V114 Lot 1 vs Prevnar 13™; Type 9V; Test type: Other; GMC Ratio = 0.88, 95% CI 2-sided [0.77 to 1.00] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 9: Comparison: V114 Lot 1 vs Prevnar 13™; Type 14; Test type: Other; GMC Ratio = 0.88, 95% CI 2-sided [0.75 to 1.03] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 10: Comparison: V114 Lot 1 vs Prevnar 13™; Type 18C; Test type: Other; GMC Ratio = 0.75, 95% CI 2-sided [0.66 to 0.84] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 11: Comparison: V114 Lot 1 vs Prevnar 13™; Type 19A; Test type: Other; GMC Ratio = 0.82, 95% CI 2-sided [0.73 to 0.92] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 12: Comparison: V114 Lot 1 vs Prevnar 13™; Type 19F; Test type: Other; GMC Ratio = 0.88, 95% CI 2-sided [0.79 to 0.98] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: V114 Lot 1 vs Prevnar 13™; Type 23F; Test type: Other; GMC Ratio = 0.98, 95% CI 2-sided [0.84 to 1.13] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 14: Comparison: V114 Lot 1 vs Prevnar 13™; Type 22F; Test type: Other; GMC Ratio = 92.05, 95% CI 2-sided [80.84 to 104.81] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 15: Comparison: V114 Lot 1 vs Prevnar 13™; Type 33F; Test type: Other; GMC Ratio = 34.41, 95% CI 2-sided [28.50 to 41.54] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 16: Comparison: V114 Lot 2 vs Prevnar 13™; Type 1; Test type: Other; GMC Ratio = 0.83, 95% CI 2-sided [0.74 to 0.94] — IgG GMC Ratio (V114 Lot 2/Prevnar 13™) based on ANOVA model with log-transformed IgG antibody responses as response variable and vaccination group as covariate
Statistical Analysis 17: Comparison: V114 Lot 2 vs Prevnar 13™; Type 3; Test type: Other; GMC Ratio = 1.93, 95% CI 2-sided [1.71 to 2.18] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 18: Comparison: V114 Lot 2 vs Prevnar 13™; Type 4; Test type: Other; GMC Ratio = 1.01, 95% CI 2-sided [0.90 to 1.14] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 19: Comparison: V114 Lot 2 vs Prevnar 13™; Type 5; Test type: Other; GMC Ratio = 0.83, 95% CI 2-sided [0.72 to 0.94] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 20: Comparison: V114 Lot 2 vs Prevnar 13™; Type 6A; Test type: Other; GMC Ratio = 0.57, 95% CI 2-sided [0.49 to 0.66] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 21: Comparison: V114 Lot 2 vs Prevnar 13™; Type 6B; Test type: Other; GMC Ratio = 0.90, 95% CI 2-sided [0.74 to 1.10] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 22: Comparison: V114 Lot 2 vs Prevnar 13™; Type 7F; Test type: Other; GMC Ratio = 0.81, 95% CI 2-sided [0.72 to 0.91] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 23: Comparison: V114 Lot 2 vs Prevnar 13™; Type 9V; Test type: Other; GMC Ratio = 1.07, 95% CI 2-sided [0.94 to 1.22] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 24: Comparison: V114 Lot 2 vs Prevnar 13™; Type 14; Test type: Other; GMC Ratio = 0.83, 95% CI 2-sided [0.71 to 0.97] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 25: Comparison: V114 Lot 2 vs Prevnar 13™; Type 18C; Test type: Other; GMC Ratio = 0.99, 95% CI 2-sided [0.88 to 1.12] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 26: Comparison: V114 Lot 2 vs Prevnar 13™; Type 19A; Test type: Other; GMC Ratio = 0.82, 95% CI 2-sided [0.73 to 0.92] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 27: Comparison: V114 Lot 2 vs Prevnar 13™; Type 19F; Test type: Other; GMC Ratio = 0.91, 95% CI 2-sided [0.81 to 1.01] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 28: Comparison: V114 Lot 2 vs Prevnar 13™; Type 23F; Test type: Other; GMC Ratio = 1.18, 95% CI 2-sided [1.01 to 1.37] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 29: Comparison: V114 Lot 2 vs Prevnar 13™; Type 22F; Test type: Other; GMC Ratio = 80.09, 95% CI 2-sided [70.30 to 91.24] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 30: Comparison: V114 Lot 2 vs Prevnar 13™; Type 33F; Test type: Other; GMC Ratio = 32.92, 95% CI 2-sided [27.25 to 39.78] — [estimate comment as in outcome 2, analysis 16]

3. Primary Outcome: Percentage of Participants Who Experience at Least 1 Adverse Event
Description: An adverse event (AE) is defined as any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The percentage of participants with one or more AEs was assessed.
Time Frame: Up to 1 month post Vaccination 4 (up to 14 months)
Population: All participants that received at least 1 vaccination and had data available for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Lot 1 | V114 Lot 2 | Prevnar 13™
Number analyzed (Participants) | 350 | 347 | 347
Percentage of Participants | 95.7 | 97.7 | 95.7
Statistical Analysis 1: Comparison: V114 Lot 1 vs Prevnar 13™; Difference in percentages calculated as V114 Lot 1 minus Prevnar 13™. Confidence intervals based on Miettinen and Nurminen method; Test type: Other; Difference in Percentages = 0.0, 95% CI 2-sided [-3.1 to 3.2]
Statistical Analysis 2: Comparison: V114 Lot 2 vs Prevnar 13™; Difference in percentages calculated as V114 Lot 2 minus Prevnar 13™. Confidence intervals based on Miettinen and Nurminen method; Test type: Other; Difference in Percentages = 2.0, 95% CI 2-sided [-0.7 to 5.0]

4. Primary Outcome: Percentage of Participants Who Discontinued From the Study Due to an Adverse Event
Description: The percentage of participants who discontinued the study because of an AE (as defined above) was assessed.
Time Frame: Up to 1 month post Vaccination 4 (up to 14 months)
Population: All participants that received at least 1 vaccination and had data available for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Lot 1 | V114 Lot 2 | Prevnar 13™
Number analyzed (Participants) | 350 | 347 | 347
Percentage of Participants | 0.3 | 0.3 | 0.0
Statistical Analysis 1: Comparison: V114 Lot 1 vs Prevnar 13™; [analysis description as in outcome 3, analysis 1]; Test type: Other; Difference in Percentages = 0.3, 95% CI 2-sided [-0.8 to 1.6]
Statistical Analysis 2: Comparison: V114 Lot 2 vs Prevnar 13™; [analysis description as in outcome 3, analysis 2]; Test type: Other; Difference in Percentages = 0.3, 95% CI 2-sided [-0.8 to 1.6]

5. Primary Outcome: Percentage of Participants With a Solicited Injection-site Adverse Event
Description: Injection-site AEs solicited on the Vaccine Report Card were redness, swelling, hard lump, and pain/tenderness. The percentage of participants with 1 or more solicited injection-site AEs was assessed.
Time Frame: Up to 14 days post any vaccination
Population: All participants that received at least 1 vaccination and had data available for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Lot 1 | V114 Lot 2 | Prevnar 13™
Number analyzed (Participants) | 350 | 347 | 347
Percentage of Participants | 76.6 | 76.7 | 70.3
Statistical Analysis 1: Comparison: V114 Lot 1 vs Prevnar 13™; Test type: Other; Difference in Percentages = 6.3, 95% CI 2-sided [-0.3 to 12.8] — Difference in percentages calculated as V114 Lot 1 minus Prevnar 13™
Statistical Analysis 2: Comparison: V114 Lot 2 vs Prevnar 13™; Test type: Other; Difference in Percentages = 6.3, 95% CI 2-sided [-0.2 to 12.9] — Difference in percentages calculated as V114 Lot 2 minus Prevnar 13™

6. Primary Outcome: Percentage of Participants With a Solicited Systemic Adverse Event
Description: Systemic AEs solicited on the Vaccine Report Card were fever, irritability, drowsiness, hive/welts, and appetite loss. The percentage of participants with 1 or more solicited systemic AEs was assessed.
Time Frame: Up to 14 days post any vaccination
Population: All participants that received at least 1 vaccination and had data available for endpoint.
Measure: Number; unit: Percentage of Participants
Arm/Group | V114 Lot 1 | V114 Lot 2 | Prevnar 13™
Number analyzed (Participants) | 350 | 347 | 347
Percentage of Participants | 90.3 | 92.2 | 89.6
Statistical Analysis 1: Comparison: V114 Lot 1 vs Prevnar 13™; Test type: Other; p = 0.772, Miettinen and Nurminen; Difference in Percentages = 0.7, 95% CI 2-sided [-3.9 to 5.2] — Difference in percentages calculated as V114 Lot 1 minus Prevnar 13™
Statistical Analysis 2: Comparison: V114 Lot 2 vs Prevnar 13™; Test type: Other; p = 0.235, Miettinen and Nurminen; Difference in Percentages = 2.6, 95% CI 2-sided [-1.7 to 7.0] — Difference in percentages calculated as V114 Lot 2 minus Prevnar 13™

7. Secondary Outcome: Geometric Mean Concentration of Serotype-specific Pneumococcal IgG Antibody for the 13 Common Serotypes in V114 and Prevnar and the 2 Serotypes Unique to V114: Pre-vaccination 4
Description: Serotype-specific pneumococcal IgG antibody was assayed using the MSD Pn electrochemiluminescence assay.
Time Frame: Before Vaccination 4 (Month 10 to 13)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 Lot 1 | V114 Lot 2 | Prevnar 13™
Number analyzed (Participants) | 329 | 330 | 332
µg/mL
  Type 1: number analyzed (Participants) | 280 | 283 | 287
  Type 1 | 0.32 [0.29 to 0.34] | 0.35 [0.33 to 0.38] | 0.46 [0.43 to 0.50]
  Type 3: number analyzed (Participants) | 280 | 283 | 287
  Type 3 | 0.25 [0.23 to 0.27] | 0.26 [0.24 to 0.29] | 0.12 [0.11 to 0.14]
  Type 4: number analyzed (Participants) | 280 | 283 | 287
  Type 4 | 0.26 [0.24 to 0.28] | 0.26 [0.24 to 0.27] | 0.27 [0.25 to 0.29]
  Type 5: number analyzed (Participants) | 280 | 283 | 287
  Type 5 | 0.74 [0.69 to 0.80] | 0.74 [0.68 to 0.79] | 0.86 [0.80 to 0.92]
  Type 6A: number analyzed (Participants) | 280 | 283 | 287
  Type 6A | 0.33 [0.30 to 0.37] | 0.38 [0.35 to 0.41] | 0.58 [0.54 to 0.64]
  Type 6B: number analyzed (Participants) | 280 | 283 | 287
  Type 6B | 0.61 [0.55 to 0.67] | 0.56 [0.51 to 0.62] | 0.50 [0.46 to 0.55]
  Type 7F: number analyzed (Participants) | 280 | 283 | 287
  Type 7F | 0.77 [0.72 to 0.83] | 0.81 [0.76 to 0.88] | 1.05 [0.98 to 1.12]
  Type 9V: number analyzed (Participants) | 280 | 283 | 287
  Type 9V | 0.40 [0.37 to 0.44] | 0.41 [0.38 to 0.44] | 0.48 [0.44 to 0.52]
  Type 14: number analyzed (Participants) | 280 | 283 | 287
  Type 14 | 1.34 [1.22 to 1.48] | 1.24 [1.12 to 1.37] | 2.03 [1.83 to 2.24]
  Type 18C: number analyzed (Participants) | 280 | 283 | 287
  Type 18C | 0.28 [0.25 to 0.30] | 0.41 [0.38 to 0.44] | 0.34 [0.32 to 0.37]
  Type 19A: number analyzed (Participants) | 280 | 283 | 287
  Type 19A | 0.40 [0.36 to 0.44] | 0.41 [0.37 to 0.45] | 0.50 [0.45 to 0.55]
  Type 19F: number analyzed (Participants) | 280 | 283 | 287
  Type 19F | 0.43 [0.39 to 0.46] | 0.47 [0.43 to 0.52] | 0.57 [0.52 to 0.63]
  Type 23F: number analyzed (Participants) | 280 | 283 | 287
  Type 23F | 0.29 [0.26 to 0.32] | 0.37 [0.33 to 0.40] | 0.32 [0.28 to 0.36]
  Type 22F: number analyzed (Participants) | 280 | 283 | 287
  Type 22F | 1.30 [1.20 to 1.40] | 1.23 [1.14 to 1.32] | 0.05 [0.04 to 0.05]
  Type 33F: number analyzed (Participants) | 280 | 283 | 286
  Type 33F | 1.01 [0.92 to 1.11] | 0.95 [0.87 to 1.04] | 0.04 [0.04 to 0.04]
Statistical Analysis 1: Comparison: V114 Lot 1 vs Prevnar 13™; Type 1; Test type: Other; GMC Ratio = 0.69, 95% CI 2-sided [0.62 to 0.76] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: V114 Lot 1 vs Prevnar 13™; Type 3; Test type: Other; GMC Ratio = 2.00, 95% CI 2-sided [1.75 to 2.28] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: V114 Lot 1 vs Prevnar 13™; Type 4; Test type: Other; GMC Ratio = 0.96, 95% CI 2-sided [0.86 to 1.07] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 4: Comparison: V114 Lot 1 vs Prevnar 13™; Type 5; Test type: Other; GMC Ratio = 0.87, 95% CI 2-sided [0.78 to 0.96] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 5: Comparison: V114 Lot 1 vs Prevnar 13™; Type 6A; Test type: Other; GMC Ratio = 0.57, 95% CI 2-sided [0.50 to 0.65] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 6: Comparison: V114 Lot 1 vs Prevnar 13™; Type 6B; Test type: Other; GMC Ratio = 1.21, 95% CI 2-sided [1.06 to 1.39] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 7: Comparison: V114 Lot 1 vs Prevnar 13™; Type 7F; Test type: Other; GMC Ratio = 0.74, 95% CI 2-sided [0.67 to 0.82] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 8: Comparison: V114 Lot 1 vs Prevnar 13™; Type 9V; Test type: Other; GMC Ratio = 0.84, 95% CI 2-sided [0.74 to 0.95] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 9: Comparison: V114 Lot 1 vs Prevnar 13™; Type 14; Test type: Other; GMC Ratio = 0.66, 95% CI 2-sided [0.58 to 0.76] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 10: Comparison: V114 Lot 1 vs Prevnar 13™; Type 18C; Test type: Other; GMC Ratio = 0.80, 95% CI 2-sided [0.72 to 0.90]; IgG GMC Ratio (V114 Lot 1/Prevnar 13™) based on ANOVA model with log-transformed IgG antibody responses as response variable and vaccination group as covariate
Statistical Analysis 11: Comparison: V114 Lot 1 vs Prevnar 13™; Type 19A; Test type: Other; GMC Ratio = 0.79, 95% CI 2-sided [0.69 to 0.91] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 12: Comparison: V114 Lot 1 vs Prevnar 13™; Type 19F; Test type: Other; GMC Ratio = 0.74, 95% CI 2-sided [0.65 to 0.85] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 13: Comparison: V114 Lot 1 vs Prevnar 13™; Type 23F; Test type: Other; GMC Ratio = 0.92, 95% CI 2-sided [0.79 to 1.07] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 14: Comparison: V114 Lot 1 vs Prevnar 13™; type 22F; Test type: Other; GMC Ratio = 27.82, 95% CI 2-sided [24.64 to 31.40] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 15: Comparison: V114 Lot 1 vs Prevnar 13™; Type 33F; Test type: Other; GMC Ratio = 25.57, 95% CI 2-sided [22.61 to 28.92] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 16: Comparison: V114 Lot 2 vs Prevnar 13™; Type 1; Test type: Other; GMC ratio = 0.77, 95% CI 2-sided [0.69 to 0.85] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 17: Comparison: V114 Lot 2 vs Prevnar 13™; Type 3; Test type: Other; GMC Ratio = 2.10, 95% CI 2-sided [1.84 to 2.39] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 18: Comparison: V114 Lot 2 vs Prevnar 13™; Type 4; Test type: Other; GMC Ratio = 0.94, 95% CI 2-sided [0.85 to 1.05] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 19: Comparison: V114 Lot 2 vs Prevnar 13™; Type 5; Test type: Other; GMC Ratio = 0.86, 95% CI 2-sided [0.77 to 0.95] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 20: Comparison: V114 Lot 2 vs Prevnar 13™; Type 6A; Test type: Other; GMC Ratio = 0.65, 95% CI 2-sided [0.57 to 0.74] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 21: Comparison: V114 Lot 2 vs Prevnar 13™; Type 6B; Test type: Other; GMC Ratio = 1.12, 95% CI 2-sided [0.97 to 1.28] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 22: Comparison: V114 Lot 2 vs Prevnar 13™; Type 7F; Test type: Other; GMC Ratio = 0.78, 95% CI 2-sided [0.70 to 0.86] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 23: Comparison: V114 Lot 2 vs Prevnar 13™; Type 9V; Test type: Other; GMC Ratio = 0.86, 95% CI 2-sided [0.76 to 0.97] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 24: Comparison: V114 Lot 2 vs Prevnar 13™; Type 14; Test type: Other; GMC Ratio = 0.61, 95% CI 2-sided [0.53 to 0.70] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 25: Comparison: V114 Lot 2 vs Prevnar 13™; Type 18C; Test type: Other; GMC Ratio = 1.20, 95% CI 2-sided [1.07 to 1.34] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 26: Comparison: V114 Lot 2 vs Prevnar 13™; Type 19A; Test type: Other; GMC Ratio = 0.82, 95% CI 2-sided [0.71 to 0.94] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 27: Comparison: V114 Lot 2 vs Prevnar 13™; Type 19F; Test type: Other; GMC Ratio = 0.83, 95% CI 2-sided [0.73 to 0.94] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 28: Comparison: V114 Lot 2 vs Prevnar 13™; Type 23F; Test type: Other; GMC Ratio = 1.16, 95% CI 2-sided [0.99 to 1.35] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 29: Comparison: V114 Lot 2 vs Prevnar 13™; Type 22F; Test type: Other; GMC Ratio = 26.30, 95% CI 2-sided [23.31 to 29.68] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 30: Comparison: V114 Lot 2 vs Prevnar 13™; Type 33F; Test type: Other; GMC Ratio = 24.10, 95% CI 2-sided [21.32 to 27.25] — [estimate comment as in outcome 2, analysis 16]

8. Secondary Outcome: Geometric Mean Concentration of Serotype-specific Pneumococcal IgG Antibody for the 13 Common Serotypes in V114 and Prevnar and the 2 Serotypes Unique to V114: 1 Month Post Vaccination 4
Description: Serotype-specific pneumococcal IgG antibody was assayed using the MSD Pn electrochemiluminescence assay.
Time Frame: 1 month post vaccination 4 (Month 11-14)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | V114 Lot 1 | V114 Lot 2 | Prevnar 13™
Number analyzed (Participants) | 329 | 330 | 332
µg/mL
  Type 1: number analyzed (Participants) | 273 | 265 | 277
  Type 1 | 1.75 [1.60 to 1.92] | 2.00 [1.84 to 2.19] | 2.47 [2.24 to 2.72]
  Type 3: number analyzed (Participants) | 273 | 265 | 277
  Type 3 | 1.12 [1.03 to 1.22] | 1.16 [1.06 to 1.26] | 0.78 [0.71 to 0.85]
  Type 4: number analyzed (Participants) | 273 | 265 | 277
  Type 4 | 1.66 [1.49 to 1.85] | 1.53 [1.37 to 1.70] | 1.88 [1.69 to 2.10]
  Type 5: number analyzed (Participants) | 273 | 265 | 277
  Type 5 | 3.43 [3.09 to 3.80] | 3.24 [2.94 to 3.57] | 4.72 [4.27 to 5.21]
  Type 6A: number analyzed (Participants) | 273 | 265 | 277
  Type 6A | 4.97 [4.49 to 5.51] | 4.60 [4.21 to 5.04] | 6.94 [6.27 to 7.69]
  Type 6B: number analyzed (Participants) | 273 | 265 | 276
  Type 6B | 7.38 [6.68 to 8.15] | 5.74 [5.24 to 6.28] | 6.91 [6.25 to 7.63]
  Type 7F: number analyzed (Participants) | 273 | 265 | 277
  Type 7F | 4.25 [3.87 to 4.66] | 4.47 [4.07 to 4.91] | 6.29 [5.73 to 6.91]
  Type 9V: number analyzed (Participants) | 273 | 265 | 276
  Type 9V | 2.43 [2.20 to 2.69] | 2.71 [2.47 to 2.96] | 3.53 [3.20 to 3.89]
  Type 14: number analyzed (Participants) | 273 | 265 | 277
  Type 14 | 7.29 [6.54 to 8.14] | 7.01 [6.30 to 7.80] | 8.28 [7.47 to 9.19]
  Type 18C: number analyzed (Participants) | 273 | 265 | 277
  Type 18C | 2.75 [2.47 to 3.05] | 3.15 [2.88 to 3.45] | 2.94 [2.65 to 3.26]
  Type 19A: number analyzed (Participants) | 273 | 265 | 277
  Type 19A | 5.80 [5.33 to 6.31] | 5.35 [4.89 to 5.87] | 6.53 [5.93 to 7.18]
  Type 19F: number analyzed (Participants) | 273 | 265 | 277
  Type 19F | 5.29 [4.81 to 5.82] | 4.94 [4.53 to 5.39] | 5.47 [4.97 to 6.01]
  Type 23F: number analyzed (Participants) | 273 | 265 | 277
  Type 23F | 2.52 [2.25 to 2.83] | 3.12 [2.82 to 3.44] | 3.38 [3.02 to 3.78]
  Type 22F: number analyzed (Participants) | 273 | 265 | 277
  Type 22F | 8.60 [7.85 to 9.42] | 7.54 [6.91 to 8.23] | 0.06 [0.05 to 0.06]
  Type 33F: number analyzed (Participants) | 273 | 265 | 272
  Type 33F | 5.02 [4.59 to 5.49] | 4.39 [4.06 to 4.73] | 0.06 [0.05 to 0.06]
Statistical Analysis 1: Comparison: V114 Lot 1 vs Prevnar 13™; Type 1; Test type: Other; GMC Ratio = 0.71, 95% CI 2-sided [0.62 to 0.81] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 2: Comparison: V114 Lot 1 vs Prevnar 13™; Type 3; Test type: Other; GMC Ratio = 1.44, 95% CI 2-sided [1.27 to 1.63] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 3: Comparison: V114 Lot 1 vs Prevnar 13™; Type 4; Test type: Other; GMC Ratio = 0.88, 95% CI 2-sided [0.76 to 1.02] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 4: Comparison: V114 Lot 1 vs Prevnar 13™; Type 5; Test type: Other; GMC Ratio = 0.73, 95% CI 2-sided [0.63 to 0.84] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 5: Comparison: V114 Lot 1 vs Prevnar 13™; Type 6A; Test type: Other; GMC Ratio = 0.72, 95% CI 2-sided [0.62 to 0.82] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 6: Comparison: V114 Lot 1 vs Prevnar 13™; Type 6B; Test type: Other; GMC Ratio = 1.07, 95% CI 2-sided [0.93 to 1.22] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 7: Comparison: V114 Lot 1 vs Prevnar 13™; Type 7F; Test type: Other; GMC Ratio = 0.67, 95% CI 2-sided [0.59 to 0.77] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 8: Comparison: V114 Lot 1 vs Prevnar 13™; Type 9V; Test type: Other; GMC Ratio = 0.69, 95% CI 2-sided [0.60 to 0.79] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 9: Comparison: V114 Lot 1 vs Prevnar 13™; Type 14; Test type: Other; GMC Ratio = 0.88, 95% CI 2-sided [0.76 to 1.02] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 10: Comparison: V114 Lot 1 vs Prevnar 13™; Type 18C; Test type: Other; GMC Ratio = 0.93, 95% CI 2-sided [0.81 to 1.08] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 11: Comparison: V114 Lot 1 vs Prevnar 13™; Type 19A; Test type: Other; GMC Ratio = 0.89, 95% CI 2-sided [0.78 to 1.01] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 12: Comparison: V114 Lot 1 vs Prevnar 13™; Type 19F; Test type: Other; GMC Ratio = 0.97, 95% CI 2-sided [0.85 to 1.10] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 13: Comparison: V114 Lot 1 vs Prevnar 13™; Type 23F; Test type: Other; GMC Ratio = 0.75, 95% CI 2-sided [0.64 to 0.87] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 14: Comparison: V114 Lot 1 vs Prevnar 13™; Type 22F; Test type: Other; GMC Ratio = 149.69, 95% CI 2-sided [130.23 to 172.06] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 15: Comparison: V114 Lot 1 vs Prevnar 13™; Type 33F; Test type: Other; GMC Ratio = 90.35, 95% CI 2-sided [79.93 to 102.12] — [estimate comment as in outcome 2, analysis 2]
Statistical Analysis 16: Comparison: V114 Lot 2 vs Prevnar 13™; Type 1; Test type: Other; GMC Ratio = 0.81, 95% CI 2-sided [0.71 to 0.93] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 17: Comparison: V114 Lot 2 vs Prevnar 13™; Type 3; Test type: Other; GMC Ratio = 1.48, 95% CI 2-sided [1.31 to 1.68] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 18: Comparison: V114 Lot 2 vs Prevnar 13™; Type 4; Test type: Other; GMC Ratio = 0.81, 95% CI 2-sided [0.70 to 0.94] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 19: Comparison: V114 Lot 2 vs Prevnar 13™; Type 5; Test type: Other; GMC Ratio = 0.69, 95% CI 2-sided [0.60 to 0.79] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 20: Comparison: V114 Lot 2 vs Prevnar 13™; Type 6A; Test type: Other; GMC Ratio = 0.66, 95% CI 2-sided [0.58 to 0.76] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 21: Comparison: V114 Lot 2 vs Prevnar 13™; Type 6B; Test type: Other; GMC Ratio = 0.83, 95% CI 2-sided [0.72 to 0.95] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 22: Comparison: V114 Lot 2 vs Prevnar 13™; Type 7F; Test type: Other; GMC Ratio = 0.71, 95% CI 2-sided [0.62 to 0.81] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 23: Comparison: V114 Lot 2 vs Prevnar 13™; Type 9V; Test type: Other; GMC Ratio = 0.77, 95% CI 2-sided [0.67 to 0.88] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 24: Comparison: V114 Lot 2 vs Prevnar 13™; Type 14; Test type: Other; GMC Ratio = 0.85, 95% CI 2-sided [0.73 to 0.98] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 25: Comparison: V114 Lot 2 vs Prevnar 13™; Type 18C; Test type: Other; GMC Ratio = 1.07, 95% CI 2-sided [0.93 to 1.24] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 26: Comparison: V114 Lot 2 vs Prevnar 13™; Type 19A; Test type: Other; GMC Ratio = 0.82, 95% CI 2-sided [0.72 to 0.93] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 27: Comparison: V114 Lot 2 vs Prevnar 13™; Type 19F; Test type: Other; GMC Ratio = 0.90, 95% CI 2-sided [0.79 to 1.03] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 28: Comparison: V114 Lot 2 vs Prevnar 13™; Type 23F; Test type: Other; GMC Ratio = 0.92, 95% CI 2-sided [0.79 to 1.08] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 29: Comparison: V114 Lot 2 vs Prevnar 13™; Type 22F; Test type: Other; GMC Ratio = 131.23, 95% CI 2-sided [114.05 to 151.00] — [estimate comment as in outcome 2, analysis 16]
Statistical Analysis 30: Comparison: V114 Lot 2 vs Prevnar 13™; Type 33F; Test type: Other; GMC Ratio = 78.99, 95% CI 2-sided [69.82 to 89.36] — [estimate comment as in outcome 2, analysis 16]

ADVERSE EVENTS:
Time Frame: Up to approximately 1-month (28 to 42 days) post Vaccination 4 (up to 15 months)
Description: All enrolled participants that received at least 1 vaccination
Arm/Group | V114 Lot 1 | V114 Lot 2 | Prevnar 13™
All-Cause Mortality (participants affected / at risk) | 1/350 | 0/347 | 0/347
Serious Adverse Events (participants affected / at risk) | 18/350 | 19/347 | 15/347
Other Adverse Events (participants affected / at risk) | 333/350 | 337/347 | 330/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 Lot 1 (N=350) | V114 Lot 2 (N=347) | Prevnar 13™ (N=347)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Infantile colic (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Intussusception (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Leukoplakia oral (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pylorospasm (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Croup infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
H1N1 influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Haemophilus bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Burns second degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Fontanelle bulging (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Infantile spasms (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular atrophy (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obliterative bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V114 Lot 1 (N=350) | V114 Lot 2 (N=347) | Prevnar 13™ (N=347)
Diarrhoea (Gastrointestinal disorders) | 39 (54) | 44 (61) | 52 (59)
Teething (Gastrointestinal disorders) | 17 (23) | 26 (38) | 19 (22)
Vomiting (Gastrointestinal disorders) | 27 (31) | 23 (24) | 34 (45)
Injection site erythema (General disorders) | 151 (256) | 164 (280) | 153 (259)
Injection site induration (General disorders) | 117 (206) | 109 (195) | 113 (200)
Injection site pain (General disorders) | 198 (385) | 200 (393) | 162 (327)
Injection site swelling (General disorders) | 98 (157) | 100 (176) | 91 (142)
Pyrexia (General disorders) | 115 (199) | 128 (221) | 141 (252)
Nasopharyngitis (Infections and infestations) | 25 (27) | 20 (23) | 19 (22)
Otitis media (Infections and infestations) | 16 (16) | 16 (16) | 18 (18)
Upper respiratory tract infection (Infections and infestations) | 26 (27) | 24 (29) | 34 (42)
Decreased appetite (Metabolism and nutrition disorders) | 158 (303) | 175 (332) | 154 (289)
Somnolence (Nervous system disorders) | 221 (564) | 241 (661) | 233 (573)
Irritability (Psychiatric disorders) | 295 (1118) | 301 (1255) | 294 (1113)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (31) | 19 (23) | 19 (19)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 21 (28) | 15 (15) | 9 (10)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 15 (16) | 21 (29) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-15): https://cdn.clinicaltrials.gov/large-docs/72/NCT02987972/Prot_SAP_000.pdf